CLINICAL TRIAL: NCT05715580
Title: A Clinical Trial to Assess the Impact of Nursing Intervention in the Adherence to Drug Treatment and to a Healthy Lifestyle in Kidney Transplant Patients
Brief Title: Impact of Nursing Intervention in Kidney Transplant Recipients Adherence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital San Carlos, Madrid (Other)
Responsible Party: Principal Investigator, Araceli Faraldo Cabana, Investigador Principal, Hospital San Carlos, Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 22/325-EC_X
Record Dates: First submitted 2023-01-16; First posted 2023-02-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Kidney Transplant; Complications
Keywords: Kidney transplantation; Treatment adherence and compliance; Clinical trial; Health Education
MeSH Terms: conditions — Treatment Adherence and Compliance; Health Education

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): The nursing intervention will consist of providing information to the patient with a KT about the importance of following the prescribed therapeutic regimen, at the same time the information they may have about healthy lifestyle habits will be expanded, with special emphasis on those areas in which there has been detected, through the administered questionnaires, a lack of adherence.
  Interventions: Other: Nursing information with a Protocol
- Control group (Placebo Comparator): The control group will be informed of the same aspects following the usual clinical practice, which consists of providing the information in the immediate post-transplant period, and resolving any doubts that the patient may have during the subsequent time.
  Interventions: Other: Usual clinical practice

INTERVENTIONS:
Other: Nursing information with a Protocol — The nursing intervention will consist of providing information to the patient with a kidney transplant.
  To do this, a Committee of experts, made up of the 6 nurses from the kidney transplant Consultations of the Community of Madrid (Spain), will carry out an Information Protocol for adults with a kidney transplant, which will cover the healthy lifestyle habits described by the bibliography
  Arms: Intervention group
Other: Usual clinical practice — Nursing information following the usual clinical practice
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to analyse the impact of an informative nursing intervention in the adherence to drug treatment and a healthy lifestyle in kidney transplant patients and the effect of poor adherence on clinical predictors of poor kidney function.

The main question[s] it aims to answer are:

* Is it possible improve the drug adherence of kidney recipients with a nursing information intervention?
* Is it possible improve the healthy lifestyle adherence of kidney recipients with a nursing information intervention? Participants will be divided into two groups: Intervention group: in which a health education action will be carried out and Control group in which the usual clinical practice will be maintained.

DETAILED DESCRIPTION:
A controlled, multicenter, single-blind clinical trial will be carried out. For this, 3 measurements will be made, a first baseline, prior to the intervention, and another two follow-up six and twelve months after the first. Patients will be divided into two groups:

1. Intervention group: in which a health education action will be carried out through the delivery of an Information Guide for adults with a kidney transplant and the regulated explanation of each of the items it contains. It will be carried out by the nurse from the Kidney Transplant Clinic responsible for follow-up, who in turn will receive an online training session, prior to the start of recruitment, on what information to provide and how to provide it.
2. Control group in which the usual clinical practice will be maintained, which consists of providing the information in the immediate post-transplant period and resolving any doubts that the patient may have during the follow-up period.

The study will be carried out in the five existing Nursing Consultations, specific to Renal Transplantation, belonging to as many hospitals of the Public Health Network of the Community of Madrid.

Study population Those patients with a functioning kidney transplant, under follow-up by one of the nursing consultations where the research will be carried out, over 18 years of age who agree to participate and sign the informed consent will be selected. Patients monitored by the clinic whose habitual residence is in an Autonomous Community other than Madrid will be excluded, those in which the frequency of revision in the Renal Transplant Clinic is scheduled for more than 6 months, as well as those hyperimmunized pre-transplant patients (Presence of preformed antibodies >75%) and those who are not trained to give their informed consent and those who do not read or understand Spanish well.

Calculation of sample size and sampling. In order to achieve the main objective of evaluating the efficacy of an informative intervention by the nurse in the adherence of the kidney transplant recipient and according to the calculations made, starting from an adherence based on the bibliography, of 50% in both arms of the study, and to detect a change of at least 20% in it, a sample of 93 patients per arm will be needed, plus an estimated 10% of losses, which results in 102 patients per arm, 204 in total.

Given the high volume of subjects seen in each of the kidney transplant consultations throughout the year, it is expected to recruit the sample in the estimated period. For example, at the Hospital Clínico San Carlos and Hospital La Paz there are more than 600 patients under follow-up, while at Hospital Ramón y Cajal there are more than 800, and at Hospital 12 de Octubre more than 2,000, with an average of daily, in each one of the consultations, of minimum 20 visits.

An intermediate analysis will be carried out, when a third of the sample has undergone the assessment of the 6 months after the intervention, and based on the result obtained, the necessary sample will be recalculated.

This calculation has been estimated with the GRANMO v.7.12 program. Randomization To carry out the randomization, firstly, it will be stratified by hospital center. Once the stratification has been carried out, the random assignment will proceed by means of a simple randomization with a sequence of random numbers generated by means of the Excel® computer program, which uses the Mersenne Twister algorithm. To do this, a sequenced list will be generated that will contain even and other odd numbers in equal amounts, assigning the patients whose random number is even to the control group and to the intervention group if the number is odd. In this way, any person who attends the consultation, meets all the inclusion requirements and none of the exclusion requirements, will have the same probability of being assigned to one or the other group. The nurse from the Renal Transplant Clinic will be in charge and responsible for carrying out the assignment process, using the random sequence provided by the principal investigator in a sealed envelope, in such a way that the nurse in charge of the assignment will not know it until the same moment of carrying out the intervention or not.

Data collection The Renal Transplant Clinic nurses will select the subjects by consecutive sampling, from a given date, until completing the sample assigned to each of the five Nursing Clinics. This allocation will be carried out based on the number of patients under follow-up in each consultation.

Once the subjects have been selected by consecutive sampling from a given date, the nurse from the Renal Transplant Clinic, in charge of conducting the interview, will explain the objectives of the study to the study subject and obtain their written informed consent.

Subsequently, membership in the control group or intervention group will be randomized.

For biomedical data, an exhaustive review of the patient's Clinical History will be carried out. These data will be collected by an independent investigator, blind to the intervention group to which the patient belongs (control group or intervention group), both in the baseline assessment and in the measurements at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Have a kidney transplant
* Agree to participate

Exclusion Criteria:

* If the habitual residence is not in Madrid
* Those whose review frequency in the Kidney Transplant Consultation is planned for more than 6 months
* Pre-transplant hyperimmunized patients (Presence of preformed antibodies >75%)
* Those who are not qualified to give their informed consent
* Those who do not read or understand the document well Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2023-04-15 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Adherence to prescribed medication | Basal, 6 and 12 months after the basal
  Measured by the Morisky-Green test

SECONDARY OUTCOMES:
Changes in Adherence to physical exercise | Basal, 6 and 12 months after the basal
  Measured by the Brief Physical Activity Assessment tool
Changes in Adherence to healthy food | Basal, 6 and 12 months after the basal
  Measured by a questionnaire created for this study
Changes in alcohol consumption | Basal, 6 and 12 months after the basal
  Measured by CAGE test
Changes in tobacco consumption | Basal, 6 and 12 months after the basal
  Measured by IPA
Changes in Presence of emotional well-being | Basal, 6 and 12 months after the basal
  Measured by the WHO-5 test
Changes in Security / Prevention of unintentional injuries | Basal, 6 and 12 months after the basal
  Measured by a questionnaire created for this study

CONTACTS AND LOCATIONS:
Overall Officials: Araceli Faraldo Cabana, Nurse, Principal Investigator — Hospital San Carlos, Madrid
Locations (5):
- Spain (5):
  - Hospital General Universitario Gregorio Marañón, Madrid, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Memoria de Actividad de donación y trasplante renal España 2020 [Internet]. 2020. Available from: http://www.ont.es/infesp/Memorias/ACTIVIDAD DE DONACIÓN Y TRASPLANTE RENAL ESPAÑA 2020.pdf
- [Background] World Health Organization. Adherence to long-term therapies : evidence for action / [edited by Eduardo Sabaté] [Internet]. Geneva PP - Geneva: World Health Organization; Available from: https://apps.who.int/iris/handle/10665/42682
- [Background] Lopez V, Hernandez D, Gonzales M. Resultados globales del trasplante renal | Nefrología al día. Nefrol al Dia [Internet]. 2021;3:1-12. Available from: https://www.nefrologiaaldia.org/es-articulo-resultados-globales-del-trasplante-renal-58
- [Background] Foundation NK. Nutrition and Transplant [Internet]. 2022 [cited 2022 Jan 18]. Available from: https://www.kidney.org/nutrition/transplant
- [Background] Estrategia de promoción de la salud y prevención en el SNS [Internet]. Madrid; Available from: https://www.mscbs.gob.es/profesionales/saludPublica/prevPromocion/Estrategia/docs/EstrategiaPromocionSaludyPrevencionSNS.pdf
- [Background] El said SH, El Hoseiny S, El Raouf A, El Dahashan KF, Gad R, El Kader A. Lifestyle Modification among Post Renal Transplant Recipient. IOSR J Nurs Heal Sci. 2017;06(03):92-113
- [Background] Pagès-Puigdemont N, Valverde-Merino MI. Métodos para medir la adherencia terapeútica. Ars Pharm. 2018;59(3):163-72.
- [Background] CKD Group. Kidney Disease: Improving Global Outcomes (KDIGO). Kidney int. 2012;3(2013):1-150
- [Background] Tan X, Patel I, Chang J. Review of the four item Morisky Medication Adherence Scale (MMAS-4) and eight item Morisky Medication Adherence Sacle (MMAS-8). Inov Pharm. 2014;5(3):165.
- [Background] Staehr Johansen K. The use of well-being measures in primary health care - the DepCare project. 1998.
- [Background] World Health Organisation. Wellbeing Measures in Primary Health Care/ The Depcare Project. Rep a WHO Meet [Internet]. 1998;45. Available from: http://www.euro.who.int/__data/assets/pdf_file/0016/130750/E60246.pdf
- [Result] Meier-Kriesche HU, Ojo AO, Port FK, Arndorfer JA, Cibrik DM, Kaplan B. Survival improvement among patients with end-stage renal disease: trends over time for transplant recipients and wait-listed patients. J Am Soc Nephrol. 2001 Jun;12(6):1293-1296. doi: 10.1681/ASN.V1261293. PMID 11373354
- [Result] Thiruchelvam PT, Willicombe M, Hakim N, Taube D, Papalois V. Renal transplantation. BMJ. 2011 Nov 14;343:d7300. doi: 10.1136/bmj.d7300. No abstract available. PMID 22084316
- [Result] Senanayake S, Graves N, Healy H, Baboolal K, Barnett A, Sypek MP, Kularatna S. Donor Kidney Quality and Transplant Outcome: An Economic Evaluation of Contemporary Practice. Value Health. 2020 Dec;23(12):1561-1569. doi: 10.1016/j.jval.2020.07.007. Epub 2020 Sep 15. PMID 33248511
- [Result] Pascazio L, Nardone IB, Clarici A, Enzmann G, Grignetti M, Panzetta GO, Vecchiet C. Anxiety, depression and emotional profile in renal transplant recipients and healthy subjects: a comparative study. Transplant Proc. 2010 Nov;42(9):3586-90. doi: 10.1016/j.transproceed.2010.08.056. PMID 21094820
- [Result] Oniscu GC, Brown H, Forsythe JL. How great is the survival advantage of transplantation over dialysis in elderly patients? Nephrol Dial Transplant. 2004 Apr;19(4):945-51. doi: 10.1093/ndt/gfh022. PMID 15031354
- [Result] Kenawy AS, Gheith O, Al-Otaibi T, Othman N, Abo Atya H, Al-Otaibi M, Nagy MS. Medication compliance and lifestyle adherence in renal transplant recipients in Kuwait. Patient Prefer Adherence. 2019 Aug 30;13:1477-1486. doi: 10.2147/PPA.S209212. eCollection 2019. PMID 31564836
- [Result] Belaiche S, Decaudin B, Dharancy S, Noel C, Odou P, Hazzan M. Factors relevant to medication non-adherence in kidney transplant: a systematic review. Int J Clin Pharm. 2017 Jun;39(3):582-593. doi: 10.1007/s11096-017-0436-4. Epub 2017 Apr 3. PMID 28374343
- [Result] Couzi L, Moulin B, Morin MP, Albano L, Godin M, Barrou B, Alamartine E, Morelon E, Girardot-Seguin S, Mendes L, Misdrahi D, Cassuto E, Merville P. Factors predictive of medication nonadherence after renal transplantation: a French observational study. Transplantation. 2013 Jan 27;95(2):326-32. doi: 10.1097/TP.0b013e318271d7c1. PMID 23149477
- [Result] Hedayati P, Shahgholian N, Ghadami A. Nonadherence Behaviors and Some Related Factors in Kidney Transplant Recipients. Iran J Nurs Midwifery Res. 2017 Mar-Apr;22(2):97-101. doi: 10.4103/ijnmr.IJNMR_220_15. PMID 28584545
- [Result] Mathis AS. Managed care implications of improving long-term outcomes in organ transplantation. Am J Manag Care. 2015 Jan;21(1 Suppl):s24-30. PMID 25734417
- [Result] Dew MA, Dabbs AD, Myaskovsky L, Shyu S, Shellmer DA, DiMartini AF, Steel J, Unruh M, Switzer GE, Shapiro R, Greenhouse JB. Meta-analysis of medical regimen adherence outcomes in pediatric solid organ transplantation. Transplantation. 2009 Sep 15;88(5):736-46. doi: 10.1097/TP.0b013e3181b2a0e0. PMID 19741474
- [Result] Brahm MM, Manfro RC, Mello D, Cioato S, Goncalves LF. Evaluation of adherence to immunosuppressive drugs in kidney transplantation by control of medication dispensing. Transplant Proc. 2012 Oct;44(8):2391-3. doi: 10.1016/j.transproceed.2012.08.001. PMID 23026602
- [Result] Hardinger KL, Hutcherson T, Preston D, Murillo D. Influence of pill burden and drug cost on renal function after transplantation. Pharmacotherapy. 2012 May;32(5):427-32. doi: 10.1002/j.1875-9114.2012.01032.x. Epub 2012 Mar 30. PMID 22467382
- [Result] Pinsky BW, Takemoto SK, Lentine KL, Burroughs TE, Schnitzler MA, Salvalaggio PR. Transplant outcomes and economic costs associated with patient noncompliance to immunosuppression. Am J Transplant. 2009 Nov;9(11):2597-606. doi: 10.1111/j.1600-6143.2009.02798.x. PMID 19843035
- [Result] Spivey CA, Chisholm-Burns MA, Damadzadeh B, Billheimer D. Determining the effect of immunosuppressant adherence on graft failure risk among renal transplant recipients. Clin Transplant. 2014 Jan;28(1):96-104. doi: 10.1111/ctr.12283. Epub 2013 Dec 11. PMID 24329814
- [Result] Nassir BA, Dean CE, Li S, Salkowski N, Solid CA, Schnitzler MA, Snyder JJ, Kim SJ, Kasiske BL, Linzer M, Israni AK. Variation in Cost and Quality in Kidney Transplantation. Transplantation. 2015 Oct;99(10):2150-7. doi: 10.1097/TP.0000000000000721. PMID 25839707
- [Result] Hugon A, Roustit M, Lehmann A, Saint-Raymond C, Borrel E, Hilleret MN, Malvezzi P, Bedouch P, Pansu P, Allenet B. Influence of intention to adhere, beliefs and satisfaction about medicines on adherence in solid organ transplant recipients. Transplantation. 2014 Jul 27;98(2):222-8. doi: 10.1097/TP.0000000000000221. PMID 24926826
- [Result] Nowicka M, Gorska M, Nowicka Z, Edyko K, Gozdzik M, Kurnatowska I. Adherence to Pharmacotherapy and Lifestyle Recommendations Among Hemodialyzed Patients and Kidney Transplant Recipients. J Ren Nutr. 2021 Sep;31(5):503-511. doi: 10.1053/j.jrn.2020.12.006. Epub 2021 Feb 26. PMID 33642185
- [Result] Takahashi A, Hu SL, Bostom A. Physical Activity in Kidney Transplant Recipients: A Review. Am J Kidney Dis. 2018 Sep;72(3):433-443. doi: 10.1053/j.ajkd.2017.12.005. Epub 2018 Feb 23. PMID 29482935
- [Result] Ronco C, Mason G, Nayak Karopadi A, Milburn A, Hegbrant J. Healthcare systems and chronic kidney disease: putting the patient in control. Nephrol Dial Transplant. 2014 May;29(5):958-63. doi: 10.1093/ndt/gft457. Epub 2013 Nov 13. PMID 24235080
- [Result] Calella P, Hernandez-Sanchez S, Garofalo C, Ruiz JR, Carrero JJ, Bellizzi V. Exercise training in kidney transplant recipients: a systematic review. J Nephrol. 2019 Aug;32(4):567-579. doi: 10.1007/s40620-019-00583-5. Epub 2019 Jan 16. PMID 30649716
- [Result] Li Y, Pan A, Wang DD, Liu X, Dhana K, Franco OH, Kaptoge S, Di Angelantonio E, Stampfer M, Willett WC, Hu FB. Impact of Healthy Lifestyle Factors on Life Expectancies in the US Population. Circulation. 2018 Jul 24;138(4):345-355. doi: 10.1161/CIRCULATIONAHA.117.032047. PMID 29712712
- [Result] Taber DJ, Fleming JN, Fominaya CE, Gebregziabher M, Hunt KJ, Srinivas TR, Baliga PK, McGillicuddy JW, Egede LE. The Impact of Health Care Appointment Non-Adherence on Graft Outcomes in Kidney Transplantation. Am J Nephrol. 2017;45(1):91-98. doi: 10.1159/000453554. Epub 2016 Dec 2. PMID 27907919
- [Result] Lin SY, Fetzer SJ, Lee PC, Chen CH. Predicting adherence to health care recommendations using health promotion behaviours in kidney transplant recipients within 1-5 years post-transplant. J Clin Nurs. 2011 Dec;20(23-24):3313-21. doi: 10.1111/j.1365-2702.2011.03757.x. Epub 2011 Jul 13. PMID 21749509
- [Result] Totti V, Campione T, Mosconi G, Tame M, Tonioli M, Gregorini M, Scarpioni R, Storari A, Mignani R, Sella G, Bellis L, Cardillo M, Sangiorgi G. Observational Retrospective Study on Patient Lifestyle in the Pretransplantation and Post-transplantation Period in the Emilia-Romagna Region. Transplant Proc. 2020 Jun;52(5):1552-1555. doi: 10.1016/j.transproceed.2020.03.015. Epub 2020 May 10. PMID 32402457
- [Result] Totti V, Campione T, Mosconi G, Tame M, Todeschini P, Sella G, Roi GS, Spazzoli A, Angelini ML, Sangiorgi G, Giannini A, Bellis L, Nanni Costa A. Promotion of Pre- and Post-Transplant Physical Exercise in the Emilia-Romagna Region: The Network of the Program "Transplantation, Physical Activity, and Sport". Transplant Proc. 2019 Nov;51(9):2902-2905. doi: 10.1016/j.transproceed.2019.02.074. Epub 2019 Oct 9. PMID 31606183
- [Result] Van Loon E, Bernards J, Van Craenenbroeck AH, Naesens M. The Causes of Kidney Allograft Failure: More Than Alloimmunity. A Viewpoint Article. Transplantation. 2020 Feb;104(2):e46-e56. doi: 10.1097/TP.0000000000003012. PMID 32000235
- [Result] Morisky DE, Green LW, Levine DM. Concurrent and predictive validity of a self-reported measure of medication adherence. Med Care. 1986 Jan;24(1):67-74. doi: 10.1097/00005650-198601000-00007. PMID 3945130
- [Result] Perez-Escamilla B, Franco-Trigo L, Moullin JC, Martinez-Martinez F, Garcia-Corpas JP. Identification of validated questionnaires to measure adherence to pharmacological antihypertensive treatments. Patient Prefer Adherence. 2015 Apr 13;9:569-78. doi: 10.2147/PPA.S76139. eCollection 2015. PMID 25926723
- [Result] Culig J, Leppee M. From Morisky to Hill-bone; self-reports scales for measuring adherence to medication. Coll Antropol. 2014 Mar;38(1):55-62. PMID 24851597
- [Result] Marshall AL, Smith BJ, Bauman AE, Kaur S. Reliability and validity of a brief physical activity assessment for use by family doctors. Br J Sports Med. 2005 May;39(5):294-7; discussion 294-7. doi: 10.1136/bjsm.2004.013771. PMID 15849294
- [Result] Sanders-Pinheiro H, Colugnati FAB, Marsicano EO, De Geest S, Medina JOP; Adhere Brazil Consortium Group. Prevalence and correlates of non-adherence to immunosuppressants and to health behaviours in patients after kidney transplantation in Brazil - the ADHERE BRAZIL multicentre study: a cross-sectional study protocol. BMC Nephrol. 2018 Feb 20;19(1):41. doi: 10.1186/s12882-018-0840-6. PMID 29463231
- [Result] Puig Ribera A, Pena Chimenis O, Romaguera Bosch M, Duran Bellido E, Heras Tebar A, Sola Gonfaus M, Sarmiento Cruz M, Cid Cantarero A. [How to identify physical inactivity in primary care: validation of the Catalan and Spanish versions of 2 short questionnaires]. Aten Primaria. 2012 Aug;44(8):485-93. doi: 10.1016/j.aprim.2012.01.005. Epub 2012 Mar 29. Spanish. PMID 22463945
- [Result] Berben L, Denhaerynck K, Dobbels F, Engberg S, Vanhaecke J, Crespo-Leiro MG, Russell CL, De Geest S; BRIGHT study consortium. Building research initiative group: chronic illness management and adherence in transplantation (BRIGHT) study: study protocol. J Adv Nurs. 2015 Mar;71(3):642-54. doi: 10.1111/jan.12519. Epub 2014 Sep 26. PMID 25257974
- [Result] Ichimaru N, Nakazawa S, Yamanaka K, Kakuta Y, Abe T, Kaimori JY, Imamura R, Nonomura N, Takahara S. Adherence to Dietary Recommendations in Maintenance Phase Kidney Transplant Patients. Transplant Proc. 2016 Apr;48(3):890-2. doi: 10.1016/j.transproceed.2015.12.129. PMID 27234760
- [Result] Hall T, Krahn GL, Horner-Johnson W, Lamb G; Rehabilitation Research and Training Center Expert Panel on Health Measurement. Examining functional content in widely used Health-Related Quality of Life scales. Rehabil Psychol. 2011 May;56(2):94-99. doi: 10.1037/a0023054. PMID 21574727
- [Result] Neipp M, Karavul B, Jackobs S, Meyer zu Vilsendorf A, Richter N, Becker T, Schwarz A, Klempnauer J. Quality of life in adult transplant recipients more than 15 years after kidney transplantation. Transplantation. 2006 Jun 27;81(12):1640-4. doi: 10.1097/01.tp.0000226070.74443.fb. PMID 16794528
- [Result] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c332. doi: 10.1136/bmj.c332. PMID 20332509
- [Derived] Faraldo-Cabana A, Sanchez-Fructuoso A, Perez-Flores I, Beneit-Montesinos JV, Munoz-Jimenez D, Peix Jimenez B, Asensio Arredondo S, Nuno Santana EI, Santana Valeros MJ, Hidalgo Gonzalez V, Gonzalez Garcia F, Ortuno-Soriano I. Development of an Information Guideline for Kidney Transplant Recipients in a Clinical Trial: Protocol for a Modified Delphi Method. JMIR Res Protoc. 2023 Nov 6;12:e46961. doi: 10.2196/46961. PMID 37930773